CLINICAL TRIAL: NCT00777842
Title: Silencing the c-Myc Gene Using Third Generation Antisense Restenosis Therapy
Brief Title: Evaluation of the GTX™ 5126 DES Coronary Stent System in the Treatment of Patients With a Lesion in the Coronary Artery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In this feasibility study device did not perform as well as expected.
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-010; 100021, CSCT
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (1):
- 1 (Experimental): Device
  Interventions: Device: GTX™ Drug Eluting Coronary Stent System

INTERVENTIONS:
Device: GTX™ Drug Eluting Coronary Stent System — Drug eluting stent

SUMMARY:
The GTX™ Drug Eluting Coronary Stent System is intended for the treatment of patients with a lesion in the coronary artery.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has discrete de novo lesion of a coronary artery with symptomatic ischemic heart disease
* Planned treatment of one lesion with a single stent
* Denovo type A, B1 lesions with a Reference diameter between 3.0 and 3.5mm and a lesion length between 5 and 16mm

Key Exclusion Criteria:

* Diabetic (HbA1C >6.0)
* Platelet count < 100000 cells/mm3 or > 700000 cells/mm3; WBC < 3000 cells/mm3; or a hemoglobin < 10 g/dl
* Renal dysfunction with creatinine > 2.0 mg/dl
* Patient has a known pre-dilatation ejection fraction (EF) less than forty five (<45%)
* Myocardial infarction (MI) less than 3 months prior to intervention
* Patient has type B2, C lesion
* Reference artery diameter <3.0 or >3.6 mm
* Target lesion length < 5mm and >16 mm
* Other stenosis >50% in target vessel
* Known hypersensitivity or contraindication to aspirin, clopidogrel, ticlopidine, or cobalt chromium, or a sensitivity to contrast agent that, in the opinion of the investigator, cannot be adequately premedicated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Vessel Lumen Patency | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Essen, Germany